CLINICAL TRIAL: NCT05491187
Title: A Randomized Controlled Trial to Compare Between Hyperbaric Bupivacaine With and Without Fentanyl in Reducing Visceral Pain During Cesarean Delivery Under Spinal Anaesthesia in Tribhuvan University Teaching Hospital
Brief Title: Comparison Between Bupivacaine With and Without Fentanyl in Reducing Pain During Cesarean Delivery Under Spinal Anaesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Rashmi Thapa, MD Resident, Anesthesiology, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ra$@
Record Dates: First submitted 2022-08-03; First posted 2022-08-08 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Visceral Pain
MeSH Terms: conditions — Visceral Pain | interventions — Fentanyl

STUDY DESIGN:
Intervention Model Description: Participants are assigned to study where two groups of treatments B and BF are given so that one group receives only B while another group receives only BF for the duration of study.
Who Masked: Participant, Investigator
Masking Description: Patients will be randomly distributed in the two groups using computed generated numbers that will be concealed in sequentially numbered, opaque sealed envelopes.
  The envelopes will be opened by an attending nurse not involved in the study just before the procedure. The study drug will be prepared by the attending anesthesiologist/ resident who will perform the subarachnoid block. The assessment of pain and data collection, data analysis will be done by principle investigator who is blinded to procedure.
  Thus, the patients and investigating and analyzing personal will be blinded to the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B (bupivacaine group) (Active Comparator): Drug used: 0.5% hyperbaric bupivacaine heavy (8%dextrose) dose -11mg with volume of 2.2ml single administration, no repetition of intervention
  Interventions: Drug: 0.5% bupivacaine heavy
- Group BF(bupivacaine with fentanyl group) (Experimental): Drug used:- 0.5% hyperbaric bupivacaine heavy (8%dextrose) dose -10mg, 2ml and fentanyl 10mg ,0.2ml with total volume of of 2.2ml single administration, no repetition of intervention
  Interventions: Drug: 0.5% bupivacaine heavy with fentanyl

INTERVENTIONS:
Drug: 0.5% bupivacaine heavy — Spinal anesthesia with 0.5% bupivacaine heavy at L3-L4 intervertebral space using Quincke's spinal needle in sitting position, single administration for each patient
  Other Names: Anawin Heavy 0.5%
  Arms: Group B (bupivacaine group)
Drug: 0.5% bupivacaine heavy with fentanyl — Spinal anesthesia with 0.5% bupivacaine heavy with fentanyl at L3-L4 intervertebral space using Quincke's spinal needle in sitting position, single administration for each patient
  Other Names: anawin heavy 0.5% + Trofentyl
  Arms: Group BF(bupivacaine with fentanyl group)

SUMMARY:
Spinal anaesthesia with hyperbaric bupivacaine is the most commonly used anesthetic technique for cesarean section. Delivery of baby during cesarean section requires traction of peritoneum and handling of intraperitoneal organs resulting in intraoperative visceral pain. The incidence of this intraoperative visceral pain can be reduced with higher dose of hyperbaric bupivacaine (12-15mg), but increasing the dose of bupivacaine increases the risk of high sensory block resulting to major hemodynamic adverse events like hypotension, bradycardia or may lead to fetal distress. Neuraxial administration of fentanyl added to bupivacaine has been proposed to intensify the sensory block without increasing sympathetic block and also improves the quality of intraoperative analgesia thus, reduces the incidence of intraoperative visceral pain. Several studies have convincingly demonstrated efficacy of intrathecal fentanyl of different doses in improving the intraoperative analgesic effect along with its associated clinical effects. However, there has been limited research conducted to compare the analgesic effects of intrathecal fentanyl of low dose in reducing visceral pain in cesarean delivery especially in our setting.

Therefore, in this study investigator aim to compare between hyperbaric bupivacaine alone with hyperbaric bupivacaine and fentanyl in reducing the visceral pain during cesarean sectionunder spinal anaesthesia.

In this study, term parturient undergoing cesarean delivery in spinal anesthesia will be allocated in 2 groups. One group will receive intrathecal hyperbaric bupivacaine whereas another interventional group will receive hyperbaric bupivacaine with addition of fentanyl. Visceral pain will be assessed in both group using numerical pain rating scale along with monitoring of vitals. Data will be collected and will be filled up in a master chart in Microsoft Excel. Statistical analysis will be done.

DETAILED DESCRIPTION:
All the pregnant women who are planned for cesarean section will be enrolled in the study and assessed for eligibility. Patients who does not meet the inclusion criteria or those who refuse to participate will be excluded from study . Other enrolled parturient who meet the eligible criteria will be randomized and allocated to two study groups by computer generated numbers that will be concealed in sequentially numbered, opaque sealed envelopes. A day prior to surgery, eligible patients will be explained in detail about the purpose of study, need, benefits and risks of procedure. They will be instructed on the method used for sensory and motor assessments. In addition they will be explained about numerical rating scale of pain, how to use it and rate it during intraoperative period. Written informed consent will be obtained during pre anaesthetic checkup. Patients will be counselled about fasting protocol and asked to remain nil per oral of 2 hours for clear liquid, 6 hours for light foods and 8 hours for fatty food. Before surgery, premedication will be done with Tablet Pantoprazole 40 mg and Tablet Metoclopramide 10 mg at 10 pm the day before surgery and 6 am in morning of surgery. In pre-delivery room, a peripheral intravenous (IV) line will be established with 18-G IV cannula. Preloading will be done with 10 ml/kg of Lactated Ringer's solution. Baseline blood pressure, mean arterial pressure, heart rate, respiratory rate, SpO2, fetal heart rate will be recorded in pre-delivery room. In the operation theater: Standard monitor including electrocardiography, noninvasive blood pressure monitoring and pulse oximetry will be attached. Patient will be positioned in sitting position. Painting of the patient's back with 10% povidine iodine and draping with sterile drapes will be done. Identification of intervertebral space will be done and the skin will be infiltrated with lidocaine 2% under all aseptic precautions.25-gauge Quincke's spinal needle will be introduced at L3-L4 intervertebral space using a midline approach in sitting position. After ensuring free flow of cerebrospinal fluid, study drug will be given over 10 - 15 sec. Study drugs would be prepared as: In group B, Inj. 0.5% hyperbaric bupivacaine 11mg (2.2ml) will be prepared. In group BF, Inj. 0.5% hyperbaric bupivacaine 10 mg (2ml) with addition of 10mcg (0.2ml) fentanyl with total volume of 2.2 ml will be prepared. Immediately after administration of spinal anesthesia, patient will be positioned supine with wedge under right hip and the time will be recorded as "time-zero".

Fetal heart rates will be noted. Patients will receive oxygen 3L/min via nasal cannula if SpO2 decreases to <95%.NIBP and HR will be assessed every 3 minute following SAB for 15 minutes or until delivery of baby and thereafter every 5 minutes till the end of surgery. SpO2 and ECG were monitored continuously throughout the study period. Sensory level will be assessed bilaterally along the mid clavicular line using spirit soaked cotton until block reached upto T6 dermatome. Motor block will be assessed based on Modified Bromage Scale. Surgery will be allowed as soon as upper sensory level reaches T6 and Bromage scale of M3.Thereafter, the level will be checked every 2 min until maximal sensory block level is confirmed. Intra operative pain will be assessed whenever the patient complains of pain or discomfort during surgery. If somatic pain occur (at time of incision to skin or subcutaneous tissue), spinal anesthesia will be converted to general anesthesia and excluded from study. For visceral pain, patient will be asked to express the pain in Numerical Rating Scale (0-10).

Assessment of visceral pain will be mainly done during ;- Delivery of baby with fundal pressure application, exteriorization of uterus, handling of other intraperitoneal organs like bowels, adnexa so as to clear off the secretions and blood, suturing of visceral peritoneum, placement of uterus back to abdominal cavity after repair. Each time NRS is 4 or more it will be considered as inadequate analgesia and inj. Fentanyl 25 mcg will be given IV bolus. Investigator will wait for 3 min for its adequate effect. If still pain persists, then the dose of fentanyl will be increased to 1 mcg/kg. After 2 doses of fentanyl, if pain still persists then Inj. Ketamine 0.5mcg/kg IV will be given. If still pain is unbearable, general anesthesia will be administered. The need to convert to general anesthesia will be noted. Following delivery of the baby, Inj. oxytocin 3 IU will be administered bolus. Continuous infusion of oxytocin drip will be given as per need after communicating with obstetrician. APGAR score of the neonate will be evaluated at 1 minute and 5 minutes.

Hypotension will be promptly treated with intravenous fluid bolus (200 ml) and Inj.

Mephentermine 6mg IV boluses, which will be repeated if necessary. If bolus dose of Mephentermine exceeds 30mg then Inj. Phenylephrine 50 mcg IV will be given. Inj. Atropine 0.6mg will be given if bradycardia occurs. If respiratory depression occur, it will be recorded and managed as -if RR ≤10 breaths /minutes then physical stimulus will be given (tapping a patient's shoulder with calling her name ). If RR is still not increased or RR ≤ 8 breaths /minutes then Inj. Nalaoxone 0.4 mg IV will be given and will be repeated after 2-3 min if necessary. Dose of Naloxone will not be exceeded 10mg/ day. Postoperatively, follow up will be done every 15 minutes if any intraoperative adverse events is noted, otherwise every 1 hourly to assess for any hemodynamic changes and adverse events related to study drug upto 6 hours. Then, monitoring of vitals, urine output and pain management will be done upto 18 hours.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS II
* Elective cesarean deliveries under SAB
* Age ≥18 years
* Term pregnancy ≥37 weeks of gestation
* Height ≥ 150 cm

Exclusion Criteria:

* Patients with neurological, psychiatric, cardiopulmonary, hepatorenal diseases, coagulopathy
* Patient refusal to participate
* Allergy or hypersensitivity to bupivacaine or fentanyl
* Patients with communication problem

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since the study involve only pregnant women undergoing cesarean delivery, so eligible participant will be only female.
Enrollment: 72 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
To compare the incidence of intraoperative visceral pain between two groups | Assessment of visceral pain will done intraoperatively mainly during delivery of baby, exteriorization of uterus,handling of intraperitoneal organs like bowels, adenexa,suturing of visceral peritoneum during cesarean section.
  For assessment of visceral pain, numerical pain rating scale of 0-10 is used for every patients.

SECONDARY OUTCOMES:
To compare the intraoperative systolic blood pressure, diastolic blood pressure, mean arterial pressure in millimeter of mercury between two groups. | Intraoperative period and also post operative time for upto 6 hour
  Monitoring of blood pressure will be done using standard monitor so as to monitor for occurrence of any drug induced hypotension.
To compare intraoperative heart rate in beats per minute between 2 groups | Intraoperative period and also post operative time for upto 6 hour
  Monitoring of heart rate will be done using standard monitor so as to monitor for occurrence of any drug induced bradycardia
To compare intraoperative oxygen saturation (SpO2) between 2 groups | Intraoperative period and also post operative time for upto 6 hour
  Monitoring of SpO2 will be done using standard monitor so as to monitor for occurrence of respiratory depression or fall in oxygen saturation.
To compare the incidence of side effects like nausea, vomiting, respiratory depression, level of sedation, pruritus between two groups | Intraoperative period and also post operative time for upto 6 hour
  Pasero Opioid - Induced Sedation Scale (POSS) will be used for assessment of level of sedation. This score consist of :
  S Sleepy, easy to arouse
  1. Awake and alert
  2. Slightly drowsy, easily arousable
  3. Frequently drowsy, arousable, drift off to sleep during conversation
  4. Somnolent, minimal or no response to verbal or physical stimulation
  A POSS score of S, 1, or 2 indicates an acceptable level of sedation, whereas a score of 3 or 4 indicates over-sedation and the need for a reversal agent.
To assess the APGAR score of baby | Observed within 1 and 5 minute after delivery of baby
  APGAR stands for Appearance , Pulse, Grimace ,Respiratory effort ,Activity .Each category is scored with 0, 1, or 2, depending on the observed condition. It is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7, 8, or 9 is normal and is a sign that the newborn is in good health

CONTACTS AND LOCATIONS:
Overall Officials: Biswas Pradhan, MBBS,MD FCTA, Study Chair — Manmohan Cardiothoracic Vascular and Transplant Center, Institute of Medicine,TU,Nepal
Locations (1):
- Tribhuvan University Teaching Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Result] Ferrarezi, W.P.P., et al., Spinal anesthesia for elective cesarean section. Bupivacaine associated with different doses of fentanyl: randomized clinical trial. Braz J Anesthesiol, 2021. 71(6): p. 642-648. 2. Gebremedhn, E., T. Belayneh, and K. Abegaz, Analgesic Effect of Intrathecal Fentanyl as an Adjuvant to Spinal Anaesthesia in Comparison with Spinal Anaesthesia with Bupivacaine Only for Mothers Delivered by Emergency Cesarean Section. Journal of Anesthesia & Critical Care, 2017. 7: p. 1-9. 3. Choi, D.H., H.J. Ahn, and M.H. Kim, Bupivacaine-sparing effect of fentanyl in spinal anesthesia for cesarean delivery. Reg Anesth Pain Med, 2000. 25(3): p. 240-5. 4. Uppal, V. and D.M. McKeen, Strategies for prevention of spinal-associated hypotension during Cesarean delivery: Are we paying attention? Can J Anaesth, 2017. 64(10): p. 991-996. 5. Ben-David, B., et al., Low-dose bupivacaine-fentanyl spinal anesthesia for cesarean delivery. Reg Anesth Pain Med, 2000. 25(3): p. 235-9. 6. Goma, H.M., Spinal Additives in Subarachnoid Anaesthesia for Cesarean Section. 2014: IntechOpen. 7. Sia, A.T., et al., Use of hyperbaric versus isobaric bupivacaine for spinal anaesthesia for caesarean section. Cochrane Database Syst Rev, 2013(5): p. Cd005143. 8. Shafer, S.L.R.J.P.F.P., Stoelting's pharmacology and physiology in anesthetic practice. 2015. 9. Bogra, J., N. Arora, and P. Srivastava, Synergistic effect of intrathecal fentanyl and bupivacaine in spinal anesthesia for cesarean section. BMC Anesthesiology, 2005. 5(1): p. 5. 10. Ali, M.A., et al., A double-blind randomized control trial to compare the effect of varying doses of intrathecal fentanyl on clinical efficacy and side effects in parturients undergoing cesarean section. J Anaesthesiol Clin Pharmacol, 2018. 34(2): p. 221-226. 11. Uppal, V., et al., Efficacy of Intrathecal Fentanyl for Cesarean Delivery: A Systematic Review and Meta-analysis of Randomized Controlled Trials With Trial Sequential Analysis. Anesth Analg, 2020. 130(1): p. 111-125. 12. Pedersen, H., et al., Incidence of Visceral Pain during Cesarean Section: The Effect of Varying Doses of Spinal Bupivacaine. Anesthesia & Analgesia, 1989. 69(1): p. 46-49. 13. Williamson, A. and B. Hoggart, Pain: a review of three commonly used pain rating scales. J Clin Nurs, 2005. 14(7): p. 798-804. 14. Nisbet, A.T. and F. Mooney-Cotter, Comparison of selected sedation scales for reporting opioid-induced sedation assessment. Pain Manag Nurs, 2009. 10(3): p. 154-64. 15. Acharya, B., et al., Effect of low dose bupivacaine and fentanyl during elective cesarean section under spinal anesthesia Journal of Anesthesia & Clinical Research, 2019. 10: p. 1-6. 16. Edwards, R.R., Chapter 5 - Pain Assessment, in Essentials of Pain Medicine and Regional Anesthesia (Second Edition), H.T. Benzon, et al., Editors. 2005, Churchill Livingstone: Philadelphia. p. 29-34. 17. Pasero, C., Assessment of sedation during opioid administration for pain management. J Perianesth Nurs, 2009. 24(3): p. 186-90. 18. Caughey, A.B., et al., Guidelines for intraoperative care in cesarean delivery: Enhanced Recovery After Surgery Society Recommendations (Part 2). Am J Obstet Gynecol, 2018. 219(6): p. 533-544.
- See also: Bupivacaine-sparing effect of fentanyl in spinal anesthesia for cesarean delivery, In 2000, Choi et al.published double blinded, prospective study involving 120 parturients undergoing cesarean delivery. — https://pubmed.ncbi.nlm.nih.gov/10834777/
- See also: Spinal anesthesia for elective cesarean section. Bupivacaine associated with different doses of fentanyl: randomized clinical trial — https://www.bjan-sba.org/article/10.1016/j.bjane.2021.03.030/pdf/rba-71-6-611fecf0a9539573ed51f022.pdf